CLINICAL TRIAL: NCT02912520
Title: Comparison of IgA Levels in the Bronchoalveolar Lavage Fluid of Patients With and Without Antibiotic Therapy
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Oliver Robak, MD, Medical University of Vienna
Other Study IDs: ORV001
Record Dates: First submitted 2016-09-13; First posted 2016-09-23 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Immunoglobulin A
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bronchoalveolar lavage fluid of patients with and without antibiotic therapy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with antibiotic therapy: Patients with antibiotic therapy for 2 weeks.
  Interventions: Drug: Anti-Bacterial Agents
- Patients without antibiotic therapy: Patients without any antibiotic therapy in the last 3 months.

INTERVENTIONS:
Drug: Anti-Bacterial Agents — administration of any antibiotic substance(s) over the course of 2 weeks
  Groups: Patients with antibiotic therapy

SUMMARY:
Investigators hypothesize that Immunoglobine (Ig) production is influenced by the microbiota of the gut. Investigators will compare microbiota-dependent Ig production in the bronchoalveolar lavage fluid of patients with and without antibiotic therapy in order to detect significant differences.

ELIGIBILITY:
Inclusion Criteria:

* endotracheal intubation
* antibiotic therapy for 2 weeks OR no antibiotic therapy for at least 3 months

Exclusion Criteria:

* active infection
* pregnancy
* immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive inclusion of eligible patients admitted to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04-23 (Actual); Study Completion 2017-04-23 (Actual)

PRIMARY OUTCOMES:
IgA levels in the bronchoalveolar lavage fluid | 2 weeks of ICU stay

SECONDARY OUTCOMES:
number of detected bacterial, viral, and fungal infections per patient | through study completion, an average of 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Robak, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoogkamp-Korstanje JA, de Koning J, Heesemann J, Festen JJ, Houtman PM, van Oyen PL. Influence of antibiotics on IgA and IgG response and persistence of Yersinia enterocolitica in patients with Yersinia-associated spondylarthropathy. Infection. 1992 Mar-Apr;20(2):53-7. doi: 10.1007/BF01711062. PMID 1582684